CLINICAL TRIAL: NCT02107742
Title: The Influence of Injection Speed on Pain During Administration of Local Anaesthetic.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013/2297C
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Needlestick Injuries
Keywords: Injections; Time factors; Pain; Healthy volunteers; Lidocaine
MeSH Terms: conditions — Needlestick Injuries; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Injection speed (Experimental): each participant receives 3 injections with the same amount of lidocaine subcutaneously on the abdomen, given over 15, 30 and 45 seconds
  Interventions: Procedure: Normal speed lidocaine injection; Procedure: Slow lidocaine injection; Procedure: Fast lidocaine injection

INTERVENTIONS:
Procedure: Normal speed lidocaine injection — 30 seconds
Procedure: Slow lidocaine injection — speed 45 seconds
Procedure: Fast lidocaine injection — speed 15 seconds

SUMMARY:
This study will investigate the influence of injection speed on pain during injection of lidocaine. It is anticipated that a longer injection time will lead to less pain for the patient during the injection. This hypothesis will be tested on healthy volunteers, who will each receive three injections with the same amount of lidocaine subcutaneously on the abdomen. The injections will be given over 15, 30 and 45 seconds. After each injection, the subject will be asked to evaluate the pain on a Visual analog scale (0-100 mm). The aim of the study is to find a simple method for pain reduction that can be used in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years

Exclusion Criteria:

* Kidney, heart or liver disease
* Eczema or psoriasis on injection site
* Neuropathy
* Regular use of painkillers
* Hypersensitivity of Lidocaine
* Pregnancy
* Diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Pain | 60 seconds
  1. Visual Analog scale 0-100 mm
  2. Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Vilhjalmur Finsen, prof md, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of Neuroscience, NTNU, Trondheim, Norway

REFERENCES:
- [Result] Tangen LF, Lundbom JS, Skarsvag TI, Wago KJ, Ballo S, Hjelseng T, Finsen V. The influence of injection speed on pain during injection of local anaesthetic. J Plast Surg Hand Surg. 2016;50(1):7-9. doi: 10.3109/2000656X.2015.1058269. Epub 2015 Sep 28. PMID 26414074